CLINICAL TRIAL: NCT05604950
Title: Sichuan Cancer Hospital & Institute
Brief Title: Surgery Versus Non-surgical Treatment for Esophageal Squamous Cell Carcinoma in Patients Older Than 70 Years
Status: Completed | Type: Observational
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCH-TS2022; No. 2020YFH0169 (Other Grant/Funding Number: the International Cooperation Projects of Science and Technology of Sichuan Province); No. 320.6750.2020-15-3 (Other Grant/Funding Number: The Wu Jieping Clinical Research Projects)
Record Dates: First submitted 2022-10-23; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophagectomy; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- S group: underwent surgical treatment.
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions
- NS group: underwent non-surgical treatment with RT and/or chemoradiotherapy.
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions

INTERVENTIONS:
Diagnostic Test: Since the data were collected retrospectively, there were no interventions — Since the data were collected retrospectively, there were no interventions

SUMMARY:
To determine whether older patients who underwent esophagectomy had better outcome survival than those who were non-surgically treated.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology confirmed ESCC,
2. Patients with esophagectomy or radiotherapy (RT)/chemotherapy (CT),
3. Age ≥ 70.

Exclusion Criteria:

1. Having other malignant tumours,
2. Missing of required data.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Data were obtained from the Sichuan Cancer Hospital & Institute Esophageal Cancer Case Management and the department of radiation oncology multicenter databases. We retrospectively analyzed esophageal squamous cell carcinoma patients who were 70 years or older, who underwent esophagectomy or radiotherapy/chemotherapy from January 2009 to December 2017. Patients were divided into two groups: surgery and non-surgery groups. We then prospectively collected data on 284 patients with esophageal squamous cell carcinoma in the Sichuan Cancer Hospital for results verification.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Selection of treatment modalities for elderly patients with oesophageal cancer | 2009.01.01-2017.12.30
  Surgical data were retrospectively collected

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozawa S, Ito E, Kazuno A, Chino O, Nakui M, Yamamoto S, Shimada H, Makuuchi H. Thoracoscopic esophagectomy while in a prone position for esophageal cancer: a preceding anterior approach method. Surg Endosc. 2013 Jan;27(1):40-7. doi: 10.1007/s00464-012-2404-3. Epub 2012 Jun 30. PMID 22752274
- [Background] Stokes A, Collins JM, Grant BF, Scamuffa RF, Hsiao CW, Johnston SS, Ammann EM, Manson JE, Preston SH. Obesity Progression Between Young Adulthood and Midlife and Incident Diabetes: A Retrospective Cohort Study of U.S. Adults. Diabetes Care. 2018 May;41(5):1025-1031. doi: 10.2337/dc17-2336. Epub 2018 Mar 5. PMID 29506982
- [Background] Reeves GK, Pirie K, Beral V, Green J, Spencer E, Bull D; Million Women Study Collaboration. Cancer incidence and mortality in relation to body mass index in the Million Women Study: cohort study. BMJ. 2007 Dec 1;335(7630):1134. doi: 10.1136/bmj.39367.495995.AE. Epub 2007 Nov 6. PMID 17986716
- [Background] Low DE, Alderson D, Cecconello I, Chang AC, Darling GE, D'Journo XB, Griffin SM, Holscher AH, Hofstetter WL, Jobe BA, Kitagawa Y, Kucharczuk JC, Law SY, Lerut TE, Maynard N, Pera M, Peters JH, Pramesh CS, Reynolds JV, Smithers BM, van Lanschot JJ. International Consensus on Standardization of Data Collection for Complications Associated With Esophagectomy: Esophagectomy Complications Consensus Group (ECCG). Ann Surg. 2015 Aug;262(2):286-94. doi: 10.1097/SLA.0000000000001098. PMID 25607756
- [Background] Clavien PA, Sanabria JR, Strasberg SM. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Surgery. 1992 May;111(5):518-26. PMID 1598671
- [Background] Cunningham SC, Kavic SM. What is a surgical complication? World J Surg. 2009 May;33(5):1099-100; author reply 1101. doi: 10.1007/s00268-008-9881-5. No abstract available. PMID 19130118
- [Background] Ji Y, Du X, Zhu W, Yang Y, Ma J, Zhang L, Li J, Tao H, Xia J, Yang H, Huang J, Bao Y, Du D, Liu D, Wang X, Li C, Yang X, Zeng M, Liu Z, Zheng W, Pu J, Chen J, Hu W, Li P, Wang J, Xu Y, Zheng X, Chen J, Wang W, Tao G, Cai J, Zhao J, Zhu J, Jiang M, Yan Y, Xu G, Bu S, Song B, Xie K, Huang S, Zheng Y, Sheng L, Lai X, Chen Y, Cheng L, Hu X, Ji W, Fang M, Kong Y, Yu X, Li H, Li R, Shi L, Shen W, Zhu C, Lv J, Huang R, He H, Chen M. Efficacy of Concurrent Chemoradiotherapy With S-1 vs Radiotherapy Alone for Older Patients With Esophageal Cancer: A Multicenter Randomized Phase 3 Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1459-1466. doi: 10.1001/jamaoncol.2021.2705. PMID 34351356
- [Background] Mohata S, Kumar HS, Sharma N, Jhakhar SL, Beniwal S, Harsh KK. Acute treatment-related toxicity in elderly patients with good performance status compared to young patients in locally advanced esophageal carcinoma treated by definitive chemoradiation: A retrospective comparative study. J Cancer Res Ther. 2020 Jan-Mar;16(1):116-119. doi: 10.4103/jcrt.JCRT_878_18. PMID 32362620
- [Background] Zhao Q, Hu G, Xiao W, Chen Y, Shen M, Tang Q, Ning X. Comparison of definitive chemoradiotherapy and radiotherapy alone in patients older than 75 years with locally advanced esophageal carcinoma: A retrospective cohort study. Medicine (Baltimore). 2017 Sep;96(35):e7920. doi: 10.1097/MD.0000000000007920. PMID 28858114
- [Background] Wang BY, Hung WH, Wu SC, Chen HC, Huang CL, Lin CH, Chen HS. Comparison Between Esophagectomy and Definitive Chemoradiotherapy in Patients With Esophageal Cancer. Ann Thorac Surg. 2019 Apr;107(4):1060-1067. doi: 10.1016/j.athoracsur.2018.11.036. Epub 2018 Dec 17. PMID 30571951
- [Background] Nomura M, Oze I, Kodaira T, Abe T, Komori A, Narita Y, Masuishi T, Taniguchi H, Kadowaki S, Ura T, Andoh M, Tachibana H, Uemura N, Tajika M, Niwa Y, Muto M, Muro K. Comparison between surgery and definitive chemoradiotherapy for patients with resectable esophageal squamous cell carcinoma: a propensity score analysis. Int J Clin Oncol. 2016 Oct;21(5):890-898. doi: 10.1007/s10147-016-0963-3. Epub 2016 Mar 15. PMID 26980212
- [Background] Kranzfelder M, Schuster T, Geinitz H, Friess H, Buchler P. Meta-analysis of neoadjuvant treatment modalities and definitive non-surgical therapy for oesophageal squamous cell cancer. Br J Surg. 2011 Jun;98(6):768-83. doi: 10.1002/bjs.7455. Epub 2011 Apr 4. PMID 21462364
- [Background] Bedenne L, Michel P, Bouche O, Milan C, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Herr JP, Paillot B, Arveux P, Bonnetain F, Binquet C. Chemoradiation followed by surgery compared with chemoradiation alone in squamous cancer of the esophagus: FFCD 9102. J Clin Oncol. 2007 Apr 1;25(10):1160-8. doi: 10.1200/JCO.2005.04.7118. PMID 17401004
- [Result] Yuan P, Xiang J, Borg M, Chen T, Lin X, Peng X, Zheng K. Analysis of lifetime death probability for major causes of death among residents in China. BMC Public Health. 2020 Jul 11;20(1):1090. doi: 10.1186/s12889-020-09201-7. PMID 32652968
- [Result] Vlacich G, Samson PP, Perkins SM, Roach MC, Parikh PJ, Bradley JD, Lockhart AC, Puri V, Meyers BF, Kozower B, Robinson CG. Treatment utilization and outcomes in elderly patients with locally advanced esophageal carcinoma: a review of the National Cancer Database. Cancer Med. 2017 Dec;6(12):2886-2896. doi: 10.1002/cam4.1250. Epub 2017 Nov 15. PMID 29139215
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Result] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008
- [Result] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Result] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868
- [Result] Rentz J, Bull D, Harpole D, Bailey S, Neumayer L, Pappas T, Krasnicka B, Henderson W, Daley J, Khuri S. Transthoracic versus transhiatal esophagectomy: a prospective study of 945 patients. J Thorac Cardiovasc Surg. 2003 May;125(5):1114-20. doi: 10.1067/mtc.2003.315. PMID 12771885